CLINICAL TRIAL: NCT02355678
Title: The Effect of Dexamethasone Versus Local Infiltration Technique on Postoperative Nausea and Vomiting After Tonsillectomy in Children: A Randomized Double-blind Clinical Trial
Brief Title: Dexamethasone Versus Local Infiltration Technique for Tonsillectomy in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Makassed General Hospital (Other)
Responsible Party: Principal Investigator, Zoher Naja, Chairperson of Anesthesia and Pain Management Department, Makassed General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201212
Record Dates: First submitted 2015-01-26; First posted 2015-02-04 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-08

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Dexamethasone; Anesthesia, General; Tonsillectomy; Tramadol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IV Dex (Experimental): dexamethasone 0.5 mg/kg IV with placebo pre-incision infiltration
  Interventions: Drug: dexamethasone; Drug: General anesthesia; Procedure: Tonsillectomy; Procedure: gastric content suction; Drug: Tramadol hydrochloride; Drug: Propacetamol hydrochloride; Drug: Paracetamol Suppository
- Infiltration (Experimental): The infiltration will be performed by the anesthetist using a 25G- 3.5cm curved needle. A total of 1.5 ml of local anesthetic mixture will be used for each tonsil. The mixture will contain: 3 ml lidocaine 2%, 3 ml lidocaine 2% with epinephrine 1/200 000, 3 ml of bupivacaine 0.5%, 0.5 ml fentanyl 50 µg ml-1, and 0.3 ml clonidine 150 µg ml-1
  Interventions: Drug: Local anesthetic infiltration; Drug: General anesthesia; Procedure: Tonsillectomy; Procedure: gastric content suction; Drug: Tramadol hydrochloride; Drug: Propacetamol hydrochloride; Drug: Paracetamol Suppository

INTERVENTIONS:
Drug: dexamethasone — IV 0.5 mg/kg
  Arms: IV Dex
Drug: Local anesthetic infiltration — Using 25 G-3.5 cm curved needle
  Arms: Infiltration
Drug: General anesthesia — Induction by intravenous fentanyl (1.5 µg kg-1) and propofol (2.5 mg kg-1) followed by endotracheal intubation facilitated by atracurium (0.5 mg kg-1).
  Maintenance with sevoflurane 1-3%, fentanyl (1-2 µg kg-1), nitrous oxide 70% and oxygen 30%.
Procedure: Tonsillectomy — Mono-polar electrocautery or cold dissection
Procedure: gastric content suction — By orogastric tube
Drug: Tramadol hydrochloride — If Visual Analogue Scale was greater than 5
Drug: Propacetamol hydrochloride — If Visual Analogue Scale was between 4 and 5
Drug: Paracetamol Suppository — If Visual Analogue Scale was less than 4

SUMMARY:
Tonsillectomy is one of the most frequent surgical operations performed in children [1-4]. It is usually associated with postoperative nausea and vomiting (PONV) with an incidence ranging from 23% to 73% [2]. Dexamethasone has been shown to be effective in reducing PONV after tonsillectomy using standardized anesthetic technique [2, 5-7]. Previous studies utilizing a different technique, the pre-incision infiltration of local anesthesia, had shown to decrease post-tonsillectomy pain, reduce analgesic consumption and provide a rapid return to normal activity [8, 9]. Given the effectiveness of dexamethasone and the pre-incision infiltration anesthetic technique, it would be beneficial to compare the effect of each on PONV.

DETAILED DESCRIPTION:
Objective The purpose of this study is to compare the effect of dexamethasone versus the pre-incision infiltration of local anesthesia in pediatric tonsillectomy procedures. The primary outcome parameter of the study is the incidence of early PONV in the post-anesthesia care unit (PACU) and late PONV on the floor and 5 days after discharge. The secondary outcome is postoperative pain.

Methods Definitions Nausea is difficult to assess in children since they are not able to verbalize their feelings. Retching, which is the unproductive effort to vomit (no expulsion of gastric content), is considered an indicator of nausea. Therefore, for the purpose of this study, PONV is defined as vomiting and/or retching. Early PONV is defined as vomiting and/or retching in the PACU. Late PONV is defined as vomiting and/or retching on the floor and 5 days after discharge.

Study design The study will be conducted prospectively, using a randomized double-blinded placebo-controlled design. Thus, neither the surgeon nor the anesthesiologist will be aware of the injected solution content and they will not be involved in data collection. The patients and the residents who will collect the data will also be unaware of the patient's assigned group.

Sampling

Patients scheduled for total or partial tonsillectomy with or without adenoidectomy starting from January 2015, whose ages range between 2 to 13 years will be included in the study.

Exclusion criteria consisted of patients who received antiemetics, steroids, antihistaminics, or psychoactive drugs within 24 hours before surgery. Patients who are suspected to have malignant neoplasm and signs of acute pharyngeal infection will be excluded from the study. Moreover, patients who have asthma, diabetes mellitus, bleeding problems, and allergy towards bupivacaine are excluded as well.

Upon meeting the eligibility criteria and signing the consent form, patients will be allocated randomly into two equal groups using the sealed envelope method. Both groups will have general anesthesia (GA) and endotracheal intubation. Then, one group will receive dexamethasone 0.5 mg/kg IV with placebo pre-incision infiltration. The other group will receive pre-incision infiltration of 1.5 ml local anesthesia mixture in each tonsil and an equivalent volume of IV saline.

Anesthetic techniques General anesthesia General anesthesia will be induced by intravenous fentanyl (1.5 µg kg-1) and propofol (2.5 mg kg-1) followed by endotracheal intubation facilitated by atracurium (0.5 mg kg-1). Anesthesia will be subsequently maintained with sevoflurane 1-3%, fentanyl (1-2 µg kg-1), nitrous oxide 70% and oxygen 30%. The sevoflurane concentration will be adjusted with the intention of keeping the heart rate and blood pressure within 25% of pre-induction values [8, 9].

Modified infiltration technique The infiltration will be performed by the anesthetist using a 25G- 3.5cm curved needle. A total of 1.5 ml of local anesthetic mixture will be used for each tonsil. The mixture will contain: 3 ml lidocaine 2%, 3 ml lidocaine 2% with epinephrine 1/200 000, 3 ml of bupivacaine 0.5%, 0.5 ml fentanyl 50 µg ml-1, and 0.3 ml clonidine 150 µg ml-1 [8, 9].

Surgical techniques The tonsillectomy techniques were monopolar electrocautery or cold dissection. The degree of tonsillar enlargement was graded as follows: tonsils within tonsillar folds; tonsils just outside tonsillar folds; tonsils well outside tonsillar folds but not reaching uvula; tonsils reaching uvula or past uvula [3]. Towards the end of the surgery, gastric contents of all patients will be suctioned via an orogastric tube prior to extubation [10]. Patients were extubated when fully awake. Systemic IV paracetamol (15 mg/kg) was given to all patients.

Data collection Pre- and intraoperative data include: patient's demographics, surgical technique, amount of fentanyl consumed, heart rate, mean arterial pressure and oxygen concentration in addition to surgery duration. Data to be collected postoperatively in the PACU (by PACU nurse) and floor included: frequency of PONV, pain scores, antiemetic and analgesic consumption as well as patients' and surgeons' satisfaction. PONV will be assessed using questions adopted from Rhodes Index of Nausea, Vomiting and Retching (RINVR) but was modified for pediatrics [11, 12]. For children aged five years and older, pain will be measured using the Visual Analog Scale (VAS) with a score of 0 denoting no pain and 10 maximum possible pains. For children less than five years of age, the Wong-Baker faces pain scale will be used. Pain will be assessed at rest in addition to when opening the jaw, swallowing, eating soft and ordinary food. The parents will be told that they will be contacted through phone calls after their hospital discharge on a daily basis and will be asked about the pain intensity and analgesic consumption of their child. Patients will be followed-up by anesthesiology resident for five postoperative days.

Parents' satisfaction will be based on quality of communication and care provided by the anesthesiologists and nurses, in addition to parental opinion of the child's recollection and the overall experience. Surgeon satisfaction will be assessed using patients' comfort and number of phone calls made by parents.

Since the study is double-blind, neither the surgeon nor the anesthesiologist are aware of the injected solution content and were not involved in data collection. The patients and the trained nurses who collect the data are also unaware of the patient's assigned group.

Postoperative pain management For pain scores >5, 1-2 mg/kg of tramadol hydrochloride (Tramal drops, Laboratoire, Grunenthal, Aachen-Germany) would be given. If pain score is between 4 and 5, 15mg/kg intravenous propacetamol hydrochloride (Pro-Dafalgan Laboratoires, UPSA, Agen, France) will be provided. Paracetamol suppository 350 mg (Tylenol CILAG SA, Schaffhouse, Switzerland) will be administered for children with pain scores <4. Paracetamol suppository 350 mg is prescribed systematically two to four times a day as needed to all discharged children. If they experience pain with a score >5, tramadol hydrochloride will be prescribed.

Statistical Analysis Data will be statistically analyzed by chi-square test and t-test (two-tailed). P-value < 0.05 is considered significant. Results will be reported as mean and standard deviation (SD), or frequency and percentage as appropriate.

ELIGIBILITY:
Inclusion Criteria:

Patients scheduled for total or partial tonsillectomy with or without adenoidectomy

Exclusion Criteria:

Patients who received antiemetics, steroids, antihistaminics, or psychoactive drugs within 24 hours before surgery.

Patients who are suspected to have malignant neoplasm and signs of acute pharyngeal infection..

Patients who have asthma, diabetes mellitus, bleeding problems, and allergy towards bupivacaine.

Ages: 2 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 129 (Actual)
Dates: Start 2015-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative nausea and vomiting | 5 postoperative days
  incidence of early PONV in the post-anesthesia care unit (PACU) and late PONV on the floor and 5 days after discharge

SECONDARY OUTCOMES:
Postoperative pain | 5 postoperative days

CONTACTS AND LOCATIONS:
Locations (1):
- Makassed General Hospital, Beirut, Lebanon

REFERENCES:
- [Derived] Naja Z, Kanawati S, Al Khatib R, Ziade F, Naja ZZ, Naja AS, Rajab M. The effect of IV dexamethasone versus local anesthetic infiltration technique in postoperative nausea and vomiting after tonsillectomy in children: A randomized double-blind clinical trial. Int J Pediatr Otorhinolaryngol. 2017 Jan;92:21-26. doi: 10.1016/j.ijporl.2016.10.030. Epub 2016 Oct 28. PMID 28012528